CLINICAL TRIAL: NCT02307903
Title: Evaluation of Quality of Care - Haemodialysis Public-Private-Partnership, Hospital Authority (HA)
Brief Title: Evaluation of Quality of Care - Haemodialysis Public-Private-Partnership, Hospital Authority
Acronym: QoC HDPPP
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Clinical Professor, The University of Hong Kong
Other Study IDs: HKCTR-1188
Record Dates: First submitted 2013-08-28; First posted 2014-12-04 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: End-stage Renal Failure (ESRF)
Keywords: end-stage renal failure (ESRF)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- End-stage renal failure (ESRF): end-stage renal failure (ESRF)

SUMMARY:
Patients with end-stage renal failure (ESRF) have lost the function to excrete urea and maintain electrolyte balance, which is lethal unless they are given renal replacement therapy (Gibney, Hoste et al. 2008). As one of the initiatives of service improvement, the HA has introduced the haemodialysis public-private partnership (HD PPP) programme to shorten the waiting time for patients with ESRF needing HD treatment. HD PPP programme is a new service provision model that purchases healthcare services from non-Government healthcare organizations. The evaluation on the quality of care (QOC) is an essential part of the programme in order to inform future policy. The Department of Family Medicine and Primary Care of the University of Hong Kong has been appointed by the HA to carry out the evaluation of the QOC of the programme.

The Action Learning and Audit Spiral methodologies to measure whether the target standard of care intended by the HD PPP programme is achieved. Each HD PPP participating hospitals and centers will be invited to complete a structure evaluation questionnaire. Sixty patients who have agreed to join HD PPP and 60 control patients who have refused to take part in HD PPP will be included. The participants will be followed up by telephone to evaluate the effect of the programme on quality of life (QOL), patient enablement, and global rating of change in health condition. Data on the process of care and clinical outcomes of care will be retrieved from the HA medical records.

Main Outcome Measures: The primary outcomes are the proportion of participants who have received the planned process of care and adequate haemodialysis (HD) measured by the Kt/V

Data Analysis: Descriptive statistics on proportions meeting the QOC criteria will be calculated. The outcomes of HD PPP subjects will be compared at 6, 12, 24, 36 and 48 months by paired sample t-test. The outcomes between HD PPP subjects and control group will be compared by independent sample t-test or Chi-square test.

Results: The QOC of the HD PPP programme will be determined. Areas of deficiency and possible areas for quality enhancement will be identified.

Conclusion: The results of this study will provide empirical evidence on whether the HD PPP can achieve equivalent QOC as the usual HA care in order to guide service planning and policy decision making for patients with ESRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently being followed up at the HA on haemodialysis, peritoneal dialysis, or are new ESRF cases will be recruited.

Exclusion Criteria:

* Patients who do not have a good vascular access, are not hemodynamically stable for HD, are not mentally sound, ambulatory and independent, are unable to understand and communicate in Chinese language, or refuse to give consent will be excluded from the HD PPP programme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty patients currently being followed up at the HA on HD, PD, or are new ESRF cases will be recruited. Both PD and new ESRF cases must fulfill certain inclusion criterion to take part in the study. The PD patients will be enrolled into the HD PPP if they have poor ultrafiltration, inadequate dialysis, or with frequent bacterial/fungal peritonitis that failed to put back on PD; whereas new ESRF patients will be enrolled if they have previously had multiple/extensive abdominal surgeries or have any abdominal pathology that makes PD not feasible. Patients who do not have a good vascular access, are not hemodynamically stable for HD, are not mentally sound, ambulatory and independent, are unable to understand and communicate in Chinese language, or refuse to give consent will be excluded from the HD PPP programme.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2010-09; Primary Completion 2016-09 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The proportion of centers that have satisfied each of the set structure criteria. | Five years
  Interim analysis will evaluate in October, 2010; October, 2011; October, 2012; October, 2013; October, 2014
The proportion of patients who have complied with the HD PPP process of care. | Five years
  Interim analysis will evaluate in June, 2011; December, 2011; December, 2012; December, 2013; December, 2014
The proportion of patients who have adequate HD measured by the Kt/V. | Five years
  Interim analysis will evaluate in June, 2011; December, 2011, December, 2012; December, 2013; December, 2014

SECONDARY OUTCOMES:
Clinical outcomes include decompensation episodes, pre-dialysis serum calcium level, blood pressure (BP), LDL-C, patient mortality and adverse clinical events. | Five years
  Baseline, 6, 12, 24, 36, 48 months after enrolment
Patient reported outcomes (PRO) are measured by the change in Short Form -12v2 scores, the Patient ennoblement index and Global Rating of Change Scale scores | Five years
  Baseline and 6-month/12-month/24-month/36-month after the first administration of questionnaire.
Service utilization outcomes are measured by General Out-patient Clinics consultation, renal Specialist Out-patient Clinics consultation, A&E attendance rates and hospitalization rate in the past 12 months. | Five years
  Baseline and 12 months for each subject; the audit cycle will be repeated annually over a period of 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, MD, Study Chair — Department of Family Medicine and Primary Care, Faculty of Medicine, The University of Hong Kong; Julie Chen, MD, Principal Investigator — Department of Family Medicine and Primary Care, Faculity of Medicine, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong Island, Hong Kong

REFERENCES:
- [Result] Wan EY, Chen JY, Choi EP, Wong CK, Chan AK, Chan KH, Lam CL. Patterns of health-related quality of life and associated factors in Chinese patients undergoing haemodialysis. Health Qual Life Outcomes. 2015 Jul 29;13:108. doi: 10.1186/s12955-015-0308-3. PMID 26215978
- [Result] Chen JY, Choi EP, Wan EY, Chan AK, Tsang JP, Chan KH, Lo WK, Lui SL, Chu WL, Lam CL. Validation of the Disease-Specific Components of the Kidney Disease Quality of Life-36 (KDQOL-36) in Chinese Patients Undergoing Maintenance Dialysis. PLoS One. 2016 May 5;11(5):e0155188. doi: 10.1371/journal.pone.0155188. eCollection 2016. PMID 27148742
- [Result] Chen JY, Wan EY, Chan KH, Chan AK, Chan FW, Lam CL. Evaluation of the quality of care of a haemodialysis public-private partnership programme for patients with end-stage renal disease. BMC Nephrol. 2016 Jul 11;17(1):79. doi: 10.1186/s12882-016-0284-9. PMID 27401348